CLINICAL TRIAL: NCT03060317
Title: Validation of the Russian Version of Coma Recovery Scale-Revised (CRS-R)
Status: Completed | Type: Observational
Sponsor: Research Center of Neurology, Russia (Other Government)
Responsible Party: Sponsor
Other Study IDs: RusvalidCRSR
Record Dates: First submitted 2017-02-04; First posted 2017-02-23 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-03

CONDITIONS: Consciousness Disorders
Keywords: Disorders of consciousness; validation studies; coma; vegetative state
MeSH Terms: conditions — Consciousness Disorders; Coma; Persistent Vegetative State | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Validation group DOC: Examination with neurological scales.
  Interventions: Behavioral: Examination with neurological scales.

INTERVENTIONS:
Behavioral: Examination with neurological scales. — Coma Recovery Scale, Glasgo Coma Scale, FOUR scale

SUMMARY:
The purpose of this study is to validate Russian version of Coma Recovery Scale - Revised and to assess its psychometric properties.

DETAILED DESCRIPTION:
There is a need of validated scale for correct assessment for patients with disorders of consciousness (DOC) in Russia. One of the most detailed scales that provides robust results in these patients is the Coma Recovery Scale - Revised (CRS-r). The validated Russian version of CRS-r will be very helpful in clinical work and scientific research for making correct assessment of patients status and its changes over time in Russia and Russian-speaking countries.

The purpose of this study is to validate Russian version of CRS-R and to assess its psychometric properties.

The first step of the study was to perform translation of CRS-r from English into Russian according to the validation protocol:

1. Double direct translation by independent translators;
2. Combination of two Russian translations;
3. Reverse translation by native English speaker.

Final Russian version and back-translated version of the Scale were approved by the original author, Dr. J. Giacino. He approved the original validation study protocol as well.

To validate Russian version of CRS-r and to assess its psychometric properties the investigators will perform an observational study on 60 adults with disorders of consciousness of different etiology on different period of recovery after coma. It is planned to include patients with various states of consciousness (e.g., vegetative state, minimally conscious state "minus" and minimally conscious state "plus") in balanced proportions.

Every patient will be examined by two independent researchers on the same day. The patients will be examined twice with a week interval between examinations for evaluation of sensitivity of CRS-r. Test-retest reliability will be applied to investigate interrater reliability. This method will be applied as well to assess the consistency of patients' scores over time. The internal consistency of the test will be investigated by inter-rater method. For this item two researchers will conduct patient assessment with CRS-R on the same day with a small period of time between the examinations. Content validity of the test will be used for assessment of validity of CRS-R. It will be performed with expert evaluation of the content of CRS-R by the investigators. Сriterion validity will be examined by assessing the correlations of CRS-R with the scales of other questionnaires with proven high psychometric properties for consciousness disorders: the Glasgow Coma Scale and Full Outline of UnResponsiveness (FOUR) score.

ELIGIBILITY:
Inclusion Criteria:

* Adults recovering after coma in any period (persistent, permanent);
* Vegetative state or minimal conscious state;
* Locked-in syndrome.

Exclusion Criteria:

* Coma, brain death.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The group of patients will be selected from residents of Research Center of Neurology, Moscow, Russia and patients of Moscow municipal hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-07-12 (Actual); Study Completion 2017-07-12 (Actual)

PRIMARY OUTCOMES:
Coma Recovery Scale-Revised | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Piradov, PhD, Study Director — Research Center of Neurology, Moscow, Russia
Locations (1):
- Research Center of Neurology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
The investigators examine the patients with 3 scales. These original protocols could be observed by the participants after a request.

REFERENCES:
- [Background] Giacino JT, Kalmar K, Whyte J. The JFK Coma Recovery Scale-Revised: measurement characteristics and diagnostic utility. Arch Phys Med Rehabil. 2004 Dec;85(12):2020-9. doi: 10.1016/j.apmr.2004.02.033. PMID 15605342